CLINICAL TRIAL: NCT05198947
Title: Better Disease Control by Multidrug Regimen in Scabies: A Randomized Controlled Trial
Brief Title: Better Disease Control by Multidrug Regimen in Scabies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Prajwal Pandey, Assistant Professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 162/073/074-IRC
Record Dates: First submitted 2021-12-17; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Scabies
Keywords: Scabies; Permethrin; Ivermectin; Combination Regimen
MeSH Terms: conditions — Scabies | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 Permethrin only (Active Comparator): Standard regimen of permethrin 5% topical application to be repeated after 1 week.
  Interventions: Drug: Permethrin Lotion 5%
- Group 2 Permethrin and Ivermectin (Active Comparator): A combination regimen of permethrin 5% topical application with oral ivermectin 200 mcg/kg given on the single day only
  Interventions: Drug: Permethrin Lotion 5% and Oral Ivermectin 200 mcg/kg

INTERVENTIONS:
Drug: Permethrin Lotion 5% — Topical permethrin 5% lotion to apply on day 1 and repeat after 1 week.
  Arms: Group 1 Permethrin only
Drug: Permethrin Lotion 5% and Oral Ivermectin 200 mcg/kg — Topical permethrin 5% lotion and oral ivermectin 200 mcg/kg to be taken on day 1 only.
  Arms: Group 2 Permethrin and Ivermectin

SUMMARY:
Scabies is associated with significant discomfort and social taboo. Existing treatment regimen frequently fails due to lack of patient compliance. We compared single use regimen to existing standard repeat application regimen for treatment of scabies.

ELIGIBILITY:
Inclusion Criteria:

* Willing patients
* Clinical diagnosis of scabies
* Within the age limits

Exclusion Criteria:

* Unwilling patients
* Patients with severe co-morbidities requiring long term medication
* Pregnant women
* Patients who don't fulfill the age limit criteria

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Pruritus | 1 month
  Rate of relief from pruritus assessed using visual analog scale

SECONDARY OUTCOMES:
Skin lesions | 1 month
  Rate of eradication of skin lesions assessed using physician global assessment scale

CONTACTS AND LOCATIONS:
Overall Officials: Prajwal Pandey, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences; Sudha Agrawal, MD, Study Director — B.P. Koirala Institute of Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heukelbach J, Feldmeier H. Scabies. Lancet. 2006 May 27;367(9524):1767-74. doi: 10.1016/S0140-6736(06)68772-2. PMID 16731272
- [Background] FitzGerald D, Grainger RJ, Reid A. Interventions for preventing the spread of infestation in close contacts of people with scabies. Cochrane Database Syst Rev. 2014 Feb 24;2014(2):CD009943. doi: 10.1002/14651858.CD009943.pub2. PMID 24566946
- [Background] Hicks MI, Elston DM. Scabies. Dermatol Ther. 2009 Jul-Aug;22(4):279-92. doi: 10.1111/j.1529-8019.2009.01243.x. PMID 19580575
- [Background] Trettin B, Lassen JA, Andersen F, Agerskov H. The journey of having scabies-a qualitative study. J Nurs Educ Pract. 2018;9(2):1.
- [Background] Heukelbach J, Mazigo HD, Ugbomoiko US. Impact of scabies in resource-poor communities. Curr Opin Infect Dis. 2013 Apr;26(2):127-32. doi: 10.1097/QCO.0b013e32835e847b. PMID 23343887
- [Background] Strong M, Johnstone P. Interventions for treating scabies. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD000320. doi: 10.1002/14651858.CD000320.pub2. PMID 17636630
- [Background] Rosumeck S, Nast A, Dressler C. Ivermectin and permethrin for treating scabies. Cochrane Database Syst Rev. 2018 Apr 2;4(4):CD012994. doi: 10.1002/14651858.CD012994. PMID 29608022
- [Background] Mounsey KE, Holt DC, McCarthy J, Currie BJ, Walton SF. Scabies: molecular perspectives and therapeutic implications in the face of emerging drug resistance. Future Microbiol. 2008 Feb;3(1):57-66. doi: 10.2217/17460913.3.1.57. PMID 18230034
- [Background] Sunderkotter C, Aebischer A, Neufeld M, Loser C, Kreuter A, Bialek R, Hamm H, Feldmeier H. Zunahme von Skabies in Deutschland und Entwicklung resistenter Kratzemilben? Evidenz und Konsequenz. J Dtsch Dermatol Ges. 2019 Jan;17(1):15-24. doi: 10.1111/ddg.13706_g. No abstract available. PMID 30615283
- [Background] Arora P, Rudnicka L, Sar-Pomian M, Wollina U, Jafferany M, Lotti T, Sadoughifar R, Sitkowska Z, Goldust M. Scabies: A comprehensive review and current perspectives. Dermatol Ther. 2020 Jul;33(4):e13746. doi: 10.1111/dth.13746. Epub 2020 Jul 6. PMID 32484302
- [Background] Taplin D, Porcelain SL, Meinking TL, Athey RL, Chen JA, Castillero PM, Sanchez R. Community control of scabies: a model based on use of permethrin cream. Lancet. 1991 Apr 27;337(8748):1016-8. doi: 10.1016/0140-6736(91)92669-s. PMID 1673175
- [Background] Purvis RS, Tyring SK. An outbreak of lindane-resistant scabies treated successfully with permethrin 5% cream. J Am Acad Dermatol. 1991 Dec;25(6 Pt 1):1015-6. doi: 10.1016/0190-9622(91)70300-q. PMID 1725779
- [Background] 1. Mushtaq A, Khurshid K, Pal SS. Comparison of efficacy and safety of oral ivermectin with topical permethrin in treatment of scabies. J Pakistan Assoc Dermatologists. 2010;20(4):227-31.
- [Background] Sharma R, Singal A. Topical permethrin and oral ivermectin in the management of scabies: a prospective, randomized, double blind, controlled study. Indian J Dermatol Venereol Leprol. 2011 Sep-Oct;77(5):581-6. doi: 10.4103/0378-6323.84063. PMID 21860157
- [Background] Dhana A, Yen H, Okhovat JP, Cho E, Keum N, Khumalo NP. Ivermectin versus permethrin in the treatment of scabies: A systematic review and meta-analysis of randomized controlled trials. J Am Acad Dermatol. 2018 Jan;78(1):194-198. doi: 10.1016/j.jaad.2017.09.006. No abstract available. PMID 29241784
- [Background] Chhaiya SB, Patel VJ, Dave JN, Mehta DS, Shah HA. Comparative efficacy and safety of topical permethrin, topical ivermectin, and oral ivermectin in patients of uncomplicated scabies. Indian J Dermatol Venereol Leprol. 2012 Sep-Oct;78(5):605-10. doi: 10.4103/0378-6323.100571. PMID 22960817
- [Background] Goldust M, Rezaee E, Hemayat S. Treatment of scabies: Comparison of permethrin 5% versus ivermectin. J Dermatol. 2012 Jun;39(6):545-7. doi: 10.1111/j.1346-8138.2011.01481.x. Epub 2012 Mar 5. PMID 22385121
- [Background] Chandler DJ, Fuller LC. A Review of Scabies: An Infestation More than Skin Deep. Dermatology. 2019;235(2):79-90. doi: 10.1159/000495290. Epub 2018 Dec 13. PMID 30544123